CLINICAL TRIAL: NCT06056830
Title: Positron Emission Tomography Using 64Cu-SAR-bisPSMA in Participants With High-risk Prostate Cancer Prior to Radical Prostatectomy: A Prospective, Single-arm, Multi-center, Blinded-review, Phase 3 Diagnostic Performance Study
Brief Title: Positron Emission Tomography Using 64Cu-SAR-bisPSMA in Participants With High-risk Prostate Cancer Prior to Radical Prostatectomy
Acronym: CLARIFY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP04
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 64Cu-SAR-bisPSMA (Experimental): 200MBq 64Cu-SAR-bisPSMA.
  Interventions: Drug: 64Cu-SAR-bisPSMA

INTERVENTIONS:
Drug: 64Cu-SAR-bisPSMA — All Patients will receive a single administration, a bolus injection of 200MBq 64Cu-SAR-bisPSMA.

SUMMARY:
The aim for this study is to assess the diagnostic performance of 64Cu-SAR-bisPSMA PET to detect regional nodal metastases.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Signed informed consent.
* Untreated, histologically confirmed adenocarcinoma of the prostate.
* High-risk or greater PC defined by National Comprehensive Cancer Network Guidelines Version 1.202327 (clinical stage ≥T3a, or Grade Group ≥4, or PSA >20 ng/mL).
* Patients electing to undergo RP with PLND.

Exclusion Criteria:

* Administration of any high energy (>300 KeV) gamma-emitting radioisotope within 5 physical half-lives prior to Day 1.
* Known or expected hypersensitivity to 64Cu-SAR-bisPSMA or any of its components.
* Patients with known predominant small cell or neuroendocrine PC.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of 64Cu-SAR-bisPSMA PET to detect regional nodal metastases | Up to 16 weeks
  Independent primary endpoints for Day 1 and Day 2 PET: Co-primary endpoint of sensitivity and specificity of 64Cu-SAR-bisPSMA PET to detect Prostate Cancer within the pelvic lymph nodes compared to the Standard of Truth.

SECONDARY OUTCOMES:
Safety and tolerability of 64Cu-SAR-bisPSMA | Up to 16 weeks
  Incidence and severity of treatment-emergent AEs and SAEs following administration of 64Cu-SAR-bisPSMA
Consistency of 64Cu-SAR-bisPSMA PET/CT interpretations for the three central readers | Up to 16 weeks
  Inter-reader reliability of agreement estimated with a multiple-reader kappa statistic
PPV and NPV of 64Cu-SAR-bisPSMA PET to detect PC within the pelvic LNs | Up to 16 weeks
  PPV and NPV of 64Cu-SAR-bisPSMA PET to detect PC within the pelvic LNs compared to the Standard of Truth
Ability of 64Cu-SAR-bisPSMA PET to detect Prostate Cancer | Up to 16 weeks
  Sensitivity of 64Cu-SAR-bisPSMA PET to detect PC within the prostate gland compared to the Standard of Truth
Diagnostic performance of 64Cu-SAR-bisPSMA PET to detect regional nodal metastases without subregion matching | Up to 16 weeks
  Sensitivity and specificity of 64Cu-SAR-bisPSMA PET to detect PC within the pelvic LNs compared to the Standard of Truth, without the requirement of subregion (Left or Right) matching between 64Cu-SAR-bisPSMA PET and Standard of Truth

CONTACTS AND LOCATIONS:
Overall Officials: Clarity Pharmaceuticals, Study Director — Clarity Pharmaceuticals
Locations (23):
- United States (20):
  - Mayo Clinic- Phoenix, Phoenix, Arizona
  - Greater Los Angeles VA Medical Center, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Mayo Clinic- Jacksonville, Jacksonville, Florida
  - NorthShore University Health System, Glenview, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - BAMF Health, Grand Rapids, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Mayo Clinic- Rochester, Rochester, Minnesota
  - XCancer Omaha LLC, Omaha, Nebraska
  - Mount Sinai Doctors Urology Faculty Practice, New York, New York
  - Urologic Specialists, Tulsa, Oklahoma
  - Oregon Urology, Springfield, Oregon
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates of Nashville, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Urology Place, San Antonio, Texas
  - Intermountain Health, Murray, Utah
  - University of Wisconsin, Madison, Wisconsin
- Australia (3):
  - St. Vincent's Sydney, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Fiona Stanley Hospital, Murdoch, Western Australia